CLINICAL TRIAL: NCT04050085
Title: A Pilot Study of Intratumoral SD-101 (Toll-Like Receptor 9 Agonist), Nivolumab, and Radiotherapy for Treatment of Chemotherapy-Refractory Metastatic Pancreatic Adenocarcinoma
Brief Title: SD-101, Nivolumab, and Radiation Therapy in Treating Patients With Chemotherapy-Refractory Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Bristol-Myers Squibb (Industry); Dynavax Technologies Corporation (Industry)
Responsible Party: Principal Investigator, Edward Kim, Principal Investigator, University of California, Davis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1452314; NCI-2019-04928 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UCDCC#281 (Other: University of California Davis Comprehensive Cancer Center); P30CA093373 (NIH)
Record Dates: First submitted 2019-08-06; First posted 2019-08-08 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Metastatic Pancreatic Adenocarcinoma; Refractory Pancreatic Adenocarcinoma; Stage IV Pancreatic Cancer AJCC v8
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Nivolumab; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (SD-101, radiation therapy, nivolumab) (Experimental): Patients receive TLR9 agonist SD-101 intratumorally on days 1 and 8 of cycle 1 and day 1 of cycles 2-5. Treatment repeats every 2 weeks for up to 5 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo radiation therapy on days 1, 3, 5, 8, and 10 of cycle 1. Patients also receive nivolumab IV over 30 minutes on day 2. Cycles with nivolumab repeat every 2 weeks for 24 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Nivolumab; Radiation: Radiation Therapy; Drug: TLR9 Agonist SD-101

INTERVENTIONS:
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; irradiation; Radiation; Radiotherapeutics; RADIOTHERAPY; RT; Therapy, Radiation
Drug: TLR9 Agonist SD-101 — Given intratumorally
  Other Names: ISS-ODN SD-101; SD-101

SUMMARY:
This phase I trial studies the side effects of SD-101 when given together with nivolumab and radiation therapy in treating patients with pancreatic cancer that does not respond to treatment with chemotherapy (chemotherapy refractory) and has spread to other places in the body (metastatic). Drugs used in chemotherapy, such as SD-101, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Giving SD-101, nivolumab, and radiation therapy may work better in treating patients with pancreatic cancer compared to nivolumab or radiation therapy alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and tolerability of intratumoral cytidine-phospho-guanosine oligodeoxynucleotide (CpG) in combination with nivolumab and radiotherapy (RT) in chemotherapy-refractory metastatic pancreatic adenocarcinoma using Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0 criteria.

SECONDARY OBJECTIVES:

I. To obtain preliminary data on disease control rate (DCR), duration of response (DOR), progression free survival (PFS), and overall survival (OS) of intratumoral CpG in combination with nivolumab and RT in chemotherapy refractory pancreatic adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 - 2
* Able and willing to provide written informed consent
* Pathology confirmed pancreatic adenocarcinoma by histology or cytology
* Life expectancy >= 3 months
* Progression during or after greater than or equal to 1 line of systemic treatment for metastatic pancreatic adenocarcinoma. Patients who do not tolerate 1st line systemic treatment for metastatic pancreatic adenocarcinoma are also eligible
* >= 1 metastatic liver lesion amenable for radiation, intratumoral injection, and core biopsy

  * Lesion for radiation, intratumoral injection, and biopsy may not be a previously irradiated lesion but may have been previously treated with liver directed therapy (e.g., radiofrequency ablation [RFA], transarterial chemoembolization [TACE], selective internal radiation therapy [SIRT], etc.) provided there is radiographic evidence of disease progression in the interim since last local/regional treatment
* >= 1 target lesion outside the field of radiation, measurable by RECIST v1.1
* Absolute neutrophil count (ANC) >= 1000 cells/mm^3
* Platelet count >= 50,000/mm^3
* Hemoglobin >= 8 g/dL
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT) =< 5 times upper limit of normal (ULN)
* Alkaline phosphatase =< 5 times ULN
* Total bilirubin =< 2 times ULN
* Creatinine =< 2 times ULN
* Patients with hepatitis B virus are allowed if antiviral therapy has been given for > 8 weeks with viral loads < 100 IU/mL prior to the first dose of trial therapy. Subjects with hepatitis C virus are allowed. Viral loads for hepatitis B and C will be monitored every 4 weeks for patients with active hepatitis B and/or C
* Women with childbearing potential and males must be willing to use adequate birth control on trial and until 5 months for women or 7 months for men after the last of study therapy
* Ability to adhere to study schedule and protocol requirements
* Willing to undergo pre-treatment biopsy and on-treatment biopsy

Exclusion Criteria:

* Actively receiving cancer directed, systemic therapy
* Prior systemic treatment for pancreatic adenocarcinoma within 2 weeks of first study treatment
* Known active auto-immune disease or immunodeficiency requiring systemic steroid equivalent to prednisone >= 10 mg/day or immunosuppressive therapy within 14 days or 5 half-lives prior to first dose of trial therapy
* History of non-infectious pneumonitis or interstitial lung disease
* Active infection requiring systemic therapy defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment
* Pregnant or lactating women
* Live attenuated vaccine received =< 30 days before first dose of trial therapy
* Known history of positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
* Contraindications to radiotherapy including but not limited to radiation sensitivity syndromes e.g., xeroderma pigmentosum, ataxia telangiectasia
* Any significant medical condition including additional active malignancies, laboratory abnormalities, or psychiatric illness that would prevent the subject from participating and adhering to study related procedures in the view of the principal investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2022-05-14 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 30 days
  Adverse events, serious adverse events, and clinical laboratory values outside normal limits will be listed for each patient and summarized by body system and dose level in frequency tables. Severity will be graded by Common Terminology Criteria for Adverse Events version 5.0.

SECONDARY OUTCOMES:
Disease control rate | Up to 1 year
Duration of response | Up to 1 year
Progression free survival | Up to 1 year
Overall survival | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Edward J Kim, MD, PhD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Comprehensive Cancer Center, Sacramento, California, United States